CLINICAL TRIAL: NCT03464721
Title: Usability of SMART ANGEL Medical Device to Record and Transmit Health Data From Patient's Home Following Outpatient Surgery
Acronym: SMART ANGEL 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDIL/2017/PC-01; 2017-A02790-53 (Other: ANSM)
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2019-01

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery Outpatients (Experimental)
  Interventions: Device: issued with SMART ANGEL device

INTERVENTIONS:
Device: issued with SMART ANGEL device — patients will use the technology at home to record and transmit data for blood pressure and oxygen saturation

SUMMARY:
This study represents the first step for testing this device in patients in real-life situations to evaluate the technological capacities and usability by the patient

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old and less than 80 years old
* The patient is undergoing orthopedic (shoulder, foot, knee), digestive (gallbladder) or gynecological (uterus-ovary) adjustment outpatient surgery
* The patient has sufficient cognitive and intellectual ability to use the system
* The patient must undergo a training test during consultation to use the tablet and perform the measurements
* The patient must have access to 4G at home.

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant
* The patient needs emergency surgery
* The patient has a level 4 or 5 ASA psychological class
* Patient cannot have outpatient surgery for medical reasons (decompensated medical pathology), or social reasons according the the SFAR (société française anesthésie réanimation) criteria. Patient alone at home and geographically far from a hospital >30km (or >45 minutes by car).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 0
  Data collected and transmitted
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 1
  Data collected and transmitted
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 2
  Data collected and transmitted
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 3
  Data collected and transmitted
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 4
  Data collected and transmitted
Number of measures recorded using tablet for blood pressure, cardiac frequency and oxygen saturation | Day 5
  Data collected and transmitted
Concordance between data collected on tablet versus paper copies | Day 0
  Percentage correct measures
Concordance between data collected on tablet versus paper copies | Day 1
  Percentage correct measures
Concordance between data collected on tablet versus paper copies | Day 2
  Percentage correct measures
Concordance between data collected on tablet versus paper copies | Day 3
  Percentage correct measures
Concordance between data collected on tablet versus paper copies | Day 4
  Percentage correct measures
Concordance between data collected on tablet versus paper copies | Day 5
  Percentage correct measures

SECONDARY OUTCOMES:
Ease of use of medical device according to patient | Day 5
  System Usability Scale (SUS) : score 0-100
Qualitative decision-making ability from pooled results of all data from all patients | End of inclusion: Month 18
  Group of 2 experts decide whether patients should have been hospitalized, called, or left alone based on retrospective analysis of all data
Readmission rate | Month 1
  Percentage of patients readmitted to hospital
Qualitative decision-making ability from pooled results of all data from all patients on readmittance rate | End of inclusion period: Month 18
  Group of 2 experts decide whether patients should have been readmitted based on retrospective analysis of all data

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Chevallier T, Buzancais G, Occean BV, Rataboul P, Boisson C, Simon N, Lannelongue A, Chaniaud N, Gricourt Y, Lefrant JY, Cuvillon P. Feasibility of remote digital monitoring using wireless Bluetooth monitors, the Smart Angel app and an original web platform for patients following outpatient surgery: a prospective observational pilot study. BMC Anesthesiol. 2020 Oct 8;20(1):259. doi: 10.1186/s12871-020-01178-5. PMID 33032541